CLINICAL TRIAL: NCT06574659
Title: Noninvasive Ventilation Breathing Test Guiding Sequential Invasive and Noninvasive Ventilation Weaning of Patients With Acute Hypoxic Respiratory Failure: a Randomized, Multicenter, Controlled Trial
Brief Title: Noninvasive Ventilation Breathing Test Guiding Weaning in Patients With Acute Hypoxic Respiratory Failure
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: West China Hospital (Other)
Collaborators: Sichuan University (Other); Dazhou Central Hospital (Other)
Responsible Party: Principal Investigator, Kang Yan, The Chair of West China of Tian Hoapital, West China Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Huaxi ICU-NVBT
Record Dates: First submitted 2024-07-17; First posted 2024-08-28 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Acute Hypoxic Respiratory Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Assigned Interventions (Experimental): Noninvasive Ventilation Breathing Test guiding sequential invasive Ventilation and noninvasive ventilation weaning group with Ventilators.
  Interventions: Procedure: Noninvasive ventilation breathing test guiding sequential invasive Ventilation and noninvasive ventilation weaing protocol
- The standard SBT guiding weaning group (Active Comparator): The standard SBT guiding weaning protocol with Ventilators.
  Interventions: Procedure: The standard SBT guiding weaning group

INTERVENTIONS:
Procedure: Noninvasive ventilation breathing test guiding sequential invasive Ventilation and noninvasive ventilation weaing protocol — Noninvasive ventilation breathing test guiding sequential invasive Ventilation and noninvasive ventilation weaing protocol
  Arms: Assigned Interventions
Procedure: The standard SBT guiding weaning group — The standard SBT guiding weaning protocol
  Arms: The standard SBT guiding weaning group

SUMMARY:
SBT, as a routine extubation strategy for invasive mechanical ventilation, has been widely recognized. However, in recent years, studies have found that SBT may lead to delayed extubation, which has been confirmed in COPD patients but has not yet been widely accepted in patients with acute hypoxic respiratory failure. Both invasive mechanical ventilation and non-invasive mechanical ventilation are positive pressure ventilation, with the essential difference being the human-machine interface. The safe inspiratory pressure for non-invasive mechanical ventilation should not exceed 20cmH2O (1cmH2O=0.098 kPa). If the cause of respiratory failure is relieved or removed, respiratory function improves, and the patient has good airway protection ability and can tolerate non-invasive ventilation, the endotracheal tube can be removed as soon as possible to switch to non-invasive mechanical ventilation, thereby shortening the time of invasive mechanical ventilation and reducing the risk of complications. This study trial aims to identify the timing of early extubation sequential non-invasive mechanical ventilation in patients with acute hypoxic respiratory failure through non-invasive ventilation breathing tests, providing a basis for updating the process of invasive mechanical ventilation extubation.

DETAILED DESCRIPTION:
All the patients included will be randomly assigned to receive Non Invasive Ventilation Breathing Test protocol or SBT protocol.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients who have been admitted to the intensive care unit (ICU) with Acute Hypoxic Respiratory Failure. Oxygenation index less than 300mmHg, have undergone tracheal intubation, and are anticipated received invasive mechanical ventilation for more than 24 hours.

Exclusion Criteria:

* • Age over 80 years,

  * Pregnancy,
  * Consciousness disorders or intracranial hypertension caused by various reasons,
  * Neuromuscular disorders,
  * Severe cardiac dysfunction (New York Heart Association Class III or IV, acute coronary syndrome or persistent ventricular tachycardia),
  * Cardiogenic shock or after major cardiac surgery,
  * Severe liver and kidney failure,
  * Severe malnutrition,
  * Injury to the upper airway or nose and face, making it impossible to wear a nose (face) mask,
  * Severe agitation, Severe agitation, expected to be unable to cooperate with non-invasive mechanical ventilation.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-03-20 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Weaning time | From the date when the patient meets the weaning screening criteria until the date of extubation, assessed up to 28 days.
  Weaning time in hours is defined as the time period from the date when the patient meets the weaning screening criteria until the date of extubation.

SECONDARY OUTCOMES:
Arterial blood gas analysis parameters at baseline, day 1, 3, and 7 | From enrollment to Day 7.
  Arterial blood gas analysis parameters are collected at baseline, Day 1, 3, and 7, such as arterial PaO2 in mmHg.
Respiratory parameters at baseline, day 1, 3, and 7 | From enrollment to Day7.
  Respiratory parameters are collected at baseline, Day 1, 3, and 7, such as airway plateau airway pressure in cmH2O.
Hemodynamic parameters at baseline, day 1, 3, and 7 | From enrollment to Day7
  Hemodynamic parameters are collected at baseline, Day 1, 3, and 7, such as as blood pressure in mmHg.
Administration and quality of analgesia and sedation. | From enrollment until extubation, assessed up to 2 weeks.
  Administration of analgesia and sedationare collected from enrollment to days 7, such as the analgesia and sedation in ug/kg/min.
RASS scores | From enrollment until extubation, assessed up to 2 weeks.
  The RASS score is assessed using a unique measurement method, and collected from enrollment to days 7.
EIT data | From the time when patients are ready for SBT trial until 1h after extubation, assessed up to 1 week.
  Obtain EIT data for before SBT and during SBT, and during non-invasive mechanical ventilation or nasal high flow ventilation after extubation with EIT, including pulmonary ventilation indicators such as Global TV in ml.
Other outcomes: length of ICU stay and length of hospital stay | From the date of enrollment until the date of discharge, assessed up to 1 year.
  Other prognostic measures will be recorded until discharge, such as length of ICU stay and length of hospital stay in days.
Other outcomes: ICU mortality and in-hospital mortality | From the date of enrollment until the date of discharge, assessed up to 1 year.
  Other prognostic measures will be recorded until discharge, such as ICU mortality and in-hospital mortality.
Adverse events | From date of enrollment until the date of transfer out of ICU, assessed up to 3 months.
  Adverse events will be recorded from enrollment until transfer out of ICU, include the occurence rate of barotrauma, ventilator-associated pneumonia，delirium, and pressure injury on the face.

CONTACTS AND LOCATIONS:
Overall Officials: Yan Kang, Study Chair — Department of Critical Care Medicine; Yongfang Zhou, Study Chair — Department of Respiratory Care; Xiaoyi Liu, Principal Investigator — Department of Critical Care Medicine
Locations (1):
- West China Hospital,Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Yes
Any data collected during this study can be acquired from the corresponding author upon a reasonable request.
Supporting Information: CSR
Time Frame: Half a year after the publication of the research paper.
Access Criteria: Any data collected during this study can be acquired from the corresponding author upon a reasonable request.